CLINICAL TRIAL: NCT00923325
Title: A Group Wide Biology and Banking Study for Phase II Study of R1507
Brief Title: Blood and Tissue Study of Patients in NIH Protocol 08-C-0800
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090054; 09-C-0054
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2017-05-18

CONDITIONS: Sarcomas
Keywords: Biomarker Analysis; Sarcomas; Ewing's Sarcoma; Osteosarcoma; Rhabdomyosarcoma; Synovial Sarcoma; Other Sarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Ewing; Osteosarcoma; Rhabdomyosarcoma; Sarcoma, Synovial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Background:

* This study is a companion biology study to NIH protocol 08-C-0080, A Phase II Trial of R1507, a Recombinant Human Antibody to the Insulin-Like Growth Factor-1 Receptor for the Treatment of Patients with Recurrent or Refractory Ewing s Sarcoma, Osteosarcoma, Synovial Sarcoma, Rhabdomyosarcoma and Other Sarcomas.
* Analysis of tumor tissue and blood samples from patients with sarcomas who are receiving treatment with the experimental drug R1507 may help elucidate the biology of sarcomas and how they respond to certain therapies with monoclonal antibodies.

Objectives:

* To study the effect over time of R1507 on the proteins and cells in the blood and tissue of patients with sarcoma in order to learn more about how patients respond to the treatment and what changes occur in their cells.
* To discover possible new treatments for cancer.

Eligibility:

* Participants in NIH protocol 08-C-0080 for the study of R1507 to treat people with various sarcomas.

Design:

* Patients who previously agreed as part of protocol 08-C-0800 to have blood sampling for pharmacodynamic studies (blood draws to test blood for levels of R1507 and how the body affects R1507) will not have any additional blood drawn as part of this study.
* Patients who did not previously agree to pharmacodynamic sampling as part of the protocol 08-C-0800 will be asked to give 6 blood samples at various time periods during the study.
* Pathology slides or tissue blocks obtained under protocol 08-C-0800 will be forwarded to F. Hoffmann-La Roche laboratories for analysis.

DETAILED DESCRIPTION:
Background:

* R1507 is a recombinant, fully human monoclonal IgG1 antibody that binds specifically to the human IGF-1R, resulting in direct inhibition of ligand binding and loss of receptor protein on the cell surface following intracellular internalization and degradation.
* Binding of R1507 has been shown to inhibit signal transduction and proliferation and survival functions mediated by the IGF-1R in cancer cells. Pre-clinical toxicology and safety pharmacology studies have been performed with R1507 and phase 1 studies in adults have resulted in a recommended intravenous dose of 9 mg/kg weekly. Phase 1 studies are ongoing in children.
* A Phase II study (SARC011/Roche NO21157): A Phase II Trial of R1507, a Recombinant Human Antibody to the Insulin-Like Growth Factor-1 Receptor for the treatment of patients with recurrent or refractory Ewing s sarcoma, osteosarcoma, synovial sarcoma, rhabdomyosarcoma and other sarcomas will allow an opportunity to collect tumor tissue and serum samples to further characterize the biology of sarcomas and their response to IGF1-R monoclonal antibody therapy.

Objectives:

* To analyze tumor tissue for IGF-1R, phosphor (p)-IGF-1R, Akt, p-Akt, PTEN, and other candidate markers related to the mechanism of action of R1507 in the treatment of patients with sarcoma and other solid tumors.
* To determine whether specific tissue-based assays performed on diagnostic specimens will allow for the identification of newer prognostic categories and potentially new molecular targets for treatment of patients with sarcoma and other solid tumors.
* To determine whether serum levels of free IGF-I/II, total IGF-I and shed IGF-1R are of significance in the outcome of patients with sarcoma and other solid tumors.
* To identify new treatment targets for therapy. Further testing of these potential targets will be carried out in hopes of expediting translation of these findings to the clinical setting.

Eligibility:

-All patients enrolled on the Phase II study SARC011/Roche NO21157 will be eligible for enrollment.

Design:

* Unstained tumor tissue slides from samples sent for confirmatory diagnosis will be forwarded for further analysis from Central Pathology Labs in New York or Leiden to Roche Clinical Sample Operations (CSO). Tissue based assays to evaluate the status of IGF-1R downstream pathway will be performed by Roche Central Lab (HistoGeneX) and NCI Lab.
* Serum based assays of free serum IGF-I/II, total serum IGF-I and shed IGF-1R receptor will be run using the samples obtained prior to the first dose of R1507 and at specified times during treatment as described in Table 3.3. All serum samples will be shipped to the Roche CSO and forwarded for analysis to the designated laboratories. Serum based assays will be performed by Roche Central Lab (MicroCoat) and Roche Diagnostics (Penzberg).

ELIGIBILITY:
* INCLUSION CRITERIA:

All patients enrolled on the Phase II study SARC011/N021157 will be eligible for enrollment.

Signed informed consent for this study according to institutional guidelines is required.

EXCLUSION CRITERIA:

None.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-12-09; Study Completion 2017-05-18

PRIMARY OUTCOMES:
Analyze tumor tissue for markers related to the mechanism of action of R1507 | 6 months
Determine if assays will allow for better identification | 6 months
Determine whether serum levels of IGF are indicitive of patientoutcome | 6 months

SECONDARY OUTCOMES:
To determine whether specific tissue-based assays performed on diagnostic specimens will allow for the identification of newer prognostic categories and potentially new molecular targets for treatment of patients with sarcoma and other solid tum...

CONTACTS AND LOCATIONS:
Overall Officials: Lee J Helman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bonath K. [The halothane inhalation anesthesia in birds and its clinical control]. Berl Munch Tierarztl Wochenschr. 1975 Aug 1;88(15):299-301. No abstract available. German. PMID 1167146
- [Background] Myhre HO. Surgical treatment of aorto-iliac atherosclerosis. Acta Chir Scand. 1977;143(1):15-20. PMID 857553
- [Background] Rosen N, Yee D, Lippman ME, Paik S, Cullen KJ. Insulin-like growth factors in human breast cancer. Breast Cancer Res Treat. 1991 May;18 Suppl 1:S55-62. doi: 10.1007/BF02633529. PMID 1651793